CLINICAL TRIAL: NCT06482814
Title: Sleep Restriction and Parental History of Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Naima Covassin, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 24-001204; 1R01HL169320-01A1 (NIH)
Record Dates: First submitted 2024-06-26; First posted 2024-07-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Sequence AB (Experimental): Sleep restriction condition in the first period and normal sleep condition in the second period. Each period will consist of a 10-day inpatient visit comprising a 3-day/2-night baseline, followed by a 5-day/5-night experimental phase, and a 2-day/2-night recovery phase.
  Interventions: Behavioral: Partial sleep deprivation (sleep restriction); Behavioral: Normal sleep
- Study Sequence BA (Experimental): Normal sleep condition in the first period and sleep restriction condition in the second period. Each period will consist of a 10-day inpatient visit comprising a 3-day/2-night baseline, followed by a 5-day/5-night experimental phase, and a 2-day/2-night recovery phase.
  Interventions: Behavioral: Partial sleep deprivation (sleep restriction); Behavioral: Normal sleep

INTERVENTIONS:
Behavioral: Partial sleep deprivation (sleep restriction) — During the experimental segment the sleep opportunity will be restricted to 5 hours/night. During the acclimation and recovery phases a 9-hour/night sleep opportunity will be provided.
Behavioral: Normal sleep — During the normal sleep condition a 9-hour/night sleep opportunity will be provided throughout the 10-day inpatient visit.

SUMMARY:
The purpose of this study is to research the effects of partial sleep deprivation (sleep restriction) in a group of individuals whose parents have high blood pressure compared to a group of individuals whose parents have normal blood pressure.

ELIGIBILITY:
Inclusion Criteria

* Healthy adults aged 18-35 years
* Absence of any significant medical or psychiatric disease (as per the investigators' judgment)
* Nonsmoker
* Nonpregnant
* History of normal sleep duration (reported average sleep duration between 7-9 hours/night and no habitual napping)
* Hypertension status information available for both biological parents
* Ability to understand study procedures and to comply with them for the entire length of the study
* Ability to understand English and provide informed consent

Exclusion Criteria

* Age <18 or >35 years
* Body mass index <18.5 or ≥30 kg/m2
* Pregnant or lactating
* Unable to determine history of HTN in participant's biological parents or subject being adopted
* Use of tobacco, vaping, marijuana products or other drugs
* Excessive caffeine consumption (>400 mg/day)
* Excessive alcohol consumption (>7 drinks/week for women, >14 drinks/week for men)
* Office SBP/DBP ≥130/80 mmHg
* Daytime ambulatory SBP/DBP ≥130/80 mmHg
* Fasting glucose ≥126 mg/dl
* Glomerular filtration rate <60 mL/min/BSA
* History of significant medical or psychiatric disorders (as per the investigators' judgment)
* Regular use of prescription medications other than contraceptives
* Use of melatonin supplements or any other over-the-counter sleep aid
* Moderate-to-severe sleep disordered breathing (apnea/hypopnea index, AHI ≥15) or mild sleep disordered breathing (AHI 5-15) with daytime sleepiness (Epworth Sleepiness Scale >10)
* Moderate-to-severe insomnia (Insomnia Severity Index >14)
* Restless leg syndrome (as per the Cambridge-Hopkins questionnaire)
* Excessive daytime sleepiness (Epworth Sleepiness Scale >15)
* Extreme chronotype (Morningness-Eveningness Questionnaire >69 or <31)
* Night shift work
* Ongoing participation in other research studies (as per the investigators' judgment)
* Any other medical, geographic, or social factor making study participation impractical
* Not English-speaking and/or inability to provide informed consent
* Exclusionary for blood draws: hemoglobin <11.6 g/dL in women / <13.2 g/dL in men; participants with measured hemoglobin levels below these thresholds will be allowed to continue participate in study tests and procedures not involving blood draws.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
24-hour Systolic Blood Pressure (BP) | Day 2, Day 4, Day 7, and Day 9
  Systolic Blood pressure will be measured in mmHg

SECONDARY OUTCOMES:
24-hour Diastolic blood pressure (DBP) | Day 2, Day 4, Day 7, and Day 9
  Diastolic blood pressure will be measured in mmHg
Awake Systolic Blood Pressure/Diastolic Blood Pressure (SBP/DBP) | Day 2, Day 4, Day 7, and Day 9
  Awake SBP/DBP will be measured in mmHg/mmHg
Asleep Systolic Blood Pressure/Diastolic Blood Pressure (SBP/DBP) | Day 2, Day 4, Day 7, and Day 9
  Asleep SBP/DBP will be measured in mmHg/mmHg
Systolic Blood Pressure/Diastolic Blood Pressure (SBP/DBP) Nocturnal dipping | Day 2, Day 4, Day 7, and Day 9
  SBP/DBP Nocturnal dipping will be measured in percent (%)
Catecholamines | Day 2, Day 4, Day 7, and Day 9
  Catecholamines will be measured from a 24-hour urine collection.
Baroreflex Sensitivity | Day 3, Day 5, Day 8, and Day 10
  Baroreflex Sensitivity will be measured from simultaneous electrocardiography (ECG) and noninvasive beat-to-beat BP recording.
Endothelial Function | Day 3, Day 5, Day 8, and Day 10
  Endothelial function will be estimated from flow-mediated vasodilation using ultrasound.
Blood Pressure (BP) response to stressors | Day 3, Day 5, Day 8, and Day 10
  BP response to stressors will be measured in mmHg
Heart Rate response to stressors | Day 3, Day 5, Day 8, and Day 10
  Heart Rate response to stressors will be measured by ECG
DNA-methylation | Day 3, Day 5, Day 8, and Day 10
  Methylated gene markers in peripheral blood mononuclear cells will be obtained
Transcriptomic | Day 3, Day 5, Day 8, and Day 10
  Whole transcriptome in peripheral blood mononuclear cells will be obtained

OTHER OUTCOMES:
Arterial Tonometry | Day 3, Day 5, Day 8, and Day 10
  Pulse wave velocity will be measured by Applanation tonometry

CONTACTS AND LOCATIONS:
Overall Officials: Naima Covassin, Ph.D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No